CLINICAL TRIAL: NCT00000315
Title: Human Dopamine Transported Imaging in Cocaine Abuse: 1
Brief Title: Human Dopamine Transported Imaging in Cocaine Abuse: 1 - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Purpose: Treatment
Other Study IDs: NIDA-09482-1; R01-09482-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1996-11

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine

INTERVENTIONS:
Drug: Cocaine

SUMMARY:
The purpose of this study is to determine the density of DA transporters during prolonged cocaine abuse and during withdrawal from cocaine use. This aim will test the hypothesis that DA transporters are altered by cocaine abuse and reestablished during withdrawal.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-11; Study Completion 2001-12

PRIMARY OUTCOMES:
Physiological changes in: heart rate and blood pressure
Subjective effects of cocaine inducements and withdrawal
Psychological effects
Effects of investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Dean Wong, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] JNM Suppl 38(5):35P May 97.